CLINICAL TRIAL: NCT00730145
Title: A Phase I, Open-Label, Single Dose Study To Evaluate The Pharmacokinetics, Safety, And Tolerability Of PD-0332334 In Subjects Receiving Chronic Hemodialysis
Brief Title: A Single Dose Study Investigating The Elimination Of PD-0332334 In Patients Receiving Regular Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A5361032
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Renal Dialysis; Pharmacokinetics
Keywords: pharmacokinetics, PD-0332334, hemodialysis, renal dialysis
MeSH Terms: interventions — imagabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PD-0332334 (Experimental)
  Interventions: Drug: PD-0332334

INTERVENTIONS:
Drug: PD-0332334 — A single, 50 mg oral dose (2 capsules) of PD-0332334 will be administered to each hemodialysis subject
  Other Names: imagabalin

SUMMARY:
1. Quantify how much PD-0332334 is removed from the blood with hemodialysis
2. Investigate the pharmacokinetics of a single dose of PD-0332334 in subjects receiving regular hemodialysis treatments.
3. Investigate the safety and tolerability of a single dose of PD-0332334 in subjects receiving hemodialysis.

DETAILED DESCRIPTION:
Assess the elimination of PD-0332334 from the blood with hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving regular hemodialysis
* Male or female patients 18 to 65 years

Exclusion Criteria:

* Severe heart failure
* Renal transplant or renal allograft
* Illicit drug use (with the exception of prescribed sedatives)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of PD-0332334 and time of maximum plasma concentration (Tmax). Half-life of PD-0332334 in this patient population with hemodialysis and without hemodialysis | 0 to 8 days
Hemodialysis clearance of PD-0332334 from the blood, the total amount and fraction of total dose of PD-0332334 removed from the blood via hemodialysis, and the half-life of drug removal from the blood via hemodialysis | 0 to 8 days
Area under the curve (AUC) of PD-0332334 from time of study medication administration to infinity (AUCinf); AUC of PD-0332334 from time of study medication administration to last quantifiable plasma concentration (AUClast). | 0 to 8 days

SECONDARY OUTCOMES:
Assess adverse events, findings from physical examinations, clinical safety laboratory assessments, ECG, vital signs. | 0 to 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Orlando, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5361032&StudyName=A%20Single%20Dose%20Study%20Investigating%20The%20Elimination%20Of%20PD-0332334%20In%20Patients%20Receiving%20Regular%20Hemodialysis